CLINICAL TRIAL: NCT04627740
Title: A Single-Arm, Single-Center, Open-Label Pilot Study of Anti-ALPP CART-cells in Patient With Alkaline Phosphatase, Placental (ALPP)-Positive Advanced Solid Tumor
Brief Title: Anti-ALPP CAR-T Cells Immunotherapy for Advanced Solid Tumors
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Xinqiao Hospital of Chongqing (Other)
Collaborators: TCRCure Biopharma Ltd. (Industry)
Responsible Party: Principal Investigator, Qingzhu Jia, M.D., Secretary, Xinqiao Hospital of Chongqing
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: TCRCureALPPCART
Record Dates: First submitted 2020-11-05; First posted 2020-11-13 (Actual); Last update posted 2026-01-20 (Actual); Status verified 2026-01

CONDITIONS: Solid Tumors

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- CART treatment (Experimental): Cyclophosphamide will be administered at dose of 20mg/kg for 1 day and then fludarabine will be given for the next 3 days with 35mg/m2 and then the CAR-T cells will be administered
  Interventions: Drug: Retroviral vector-transduced autologous T cells to express anti-ALPP CARs

INTERVENTIONS:
Drug: Retroviral vector-transduced autologous T cells to express anti-ALPP CARs — Cyclophosphamide will be administered at dose of 20mg/kg for 1 day and then fludarabine will be given for the next 3 days with 35mg/m2 and then the CAR-T cells will be administered

SUMMARY:
The goal of this clinical trial is to evaluate the safety and efficacy of anti-ALPP chimeric antigen receptor (CAR)-modified T (CAR-T) cells in treating patients with ALPP-positive Advanced Solid Tumors.

DETAILED DESCRIPTION:
Primary Objectives:

To evaluate the number of ALPP-positive participants with treatment-related adverse events as assessed by CTCAE v4.0 after infusion with anti-ALPP CAR-T cells.

Secondary Objectives:

The number of patients experience objective response from anti-ALPP CAR-T cells treatment

To evaluate the progression-free survival (PFS) of anti-ALPP CAR-T cells in patients with ALPP-positive patients.

The number and percent of ALPP-CART cells in peripheral blood from ALPP-positive patients at 6 months after infusion

ELIGIBILITY:
Inclusion Criteria:

* Expected to survive more than 3 months
* PS 0-2
* Immunohistochemistry was confirmed to be mesothelin positive ALPP (higher than 50%)
* Patients with no curative regimen to receive
* WBC>3.5×1e+9/L,Hb>90g/L,PLT>75×1e+9/L
* HBV DNA copy number less than 100/ml
* ALT≤5ULN, AST≤5ULN, TB≤1.5ULN, ALB≥35g/L
* Understand this test and have signed informed consent

Exclusion Criteria:

* Autoimmune diseases, or any uncontrolled active disease that hinders participation in the trial
* Decompensated liver cirrhosis, liver function Child-pugh C grade
* Portal vein tumor thrombus, arterial portal fistula, hepatic arteriovenous
* Long-term use of immunosuppressive agents after organ transplantation
* Screening indicated that the target cell transfection rate was less than 30%
* Invasive pulmonary embolism, deep venous thrombosis, or other major arterial / venous thromboembolic events occurred 30 days or 30 days prior to randomization
* Subjects had an active or uncontrollable infection requiring systemic therapy 14 days or 14 days prior to randomization
* Pregnant or lactating subjects
* In the opinion of the investigator, the presence of a medical history or a history of mental state may increase the number of subjects associated with the risk factors associated with the study or study drug administration
* Subjects who have signed a written consent or who are in compliance with the study procedure; or who are unwilling or unable to comply with the study

Ages: 18 Years to 70 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 5 (Actual)
Dates: Start 2020-12-01 (Actual); Primary Completion 2025-02-28 (Actual); Study Completion 2025-08-31 (Actual)

PRIMARY OUTCOMES:
Number of patients suffering treatment-related AE | 1 year
  To evaluate the number of ALPP-positive participants with treatment-related adverse events as assessed by CTCAE v4.0 after infusion with anti-ALPP CAR-T cells.

SECONDARY OUTCOMES:
Objective response rate to ALPP-CART infusion | Eight weeks
  The number of patients experience objective response from anti-ALPP CAR-T cells treatment
Progression-free survival to ALPP-CART infusion | 6 months
  To evaluate the progression-free survival (PFS) of anti-ALPP CAR-T cells in patients with mesothelin-positive advanced ovarian carcinoma.
Number of peripheral CAR-T after infusion | 6 months
  The number of ALPP-CART cells in peripheral blood from ALPP-positive patients at 6 months after infusion

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Oncology, Xinqiao Hospital, Chongqing, Chongqing Municipality, China

IPD SHARING:
Plan to Share IPD: No